CLINICAL TRIAL: NCT01770132
Title: Open-label, Single-center, Non-randomized, Phase I, Dose-ranging Study of Endoscopic Ultrasound (EUS) Guided Photodynamic Therapy (PDT) With Photofrin® in Locally Advanced Pancreatic Cancer
Brief Title: Ultrasound-Guided Photodynamic Therapy With Photofrin & Gemcitabine for Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John DeWitt (Other)
Collaborators: American Society for Gastrointestinal Endoscopy (Other); Pinnacle Biologics Inc. (Industry)
Responsible Party: Sponsor-Investigator, John DeWitt, Principle Investigator, Indiana University
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0319; 1207009096 (Other: Indiana University Institutional Review Board)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Stage III Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dihematoporphyrin Ether; Endoscopic Ultrasound-Guided Fine Needle Aspiration; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- porfimer sodium, EUS-PDT, gemcitabine (Experimental): Patients receive porfimer sodium IV over 3-5 minutes on day 1 and undergo endoscopic ultrasonography-photodynamic therapy (EUS-PDT) on days 1, 3, 8, and 21. After completion of EUS-PDT, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 of courses 1 and 2 and on day 22 of courses 3 and 5. During courses 1-5, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After course 5, treatment with gemcitabine hydrochloride repeats every 2 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: porfimer sodium; Procedure: endoscopic ultrasonography; Procedure: photodynamic therapy; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: porfimer sodium — Given IV
  Other Names: Photofrin; Photofrin II; Porfimer
Procedure: endoscopic ultrasonography — Undergo EUS-PDT
  Other Names: endoscopic ultrasound; EUS
Procedure: photodynamic therapy — Undergo EUS-PDT
  Other Names: Light Infusion Therapy; PDT; therapy, photodynamic
Drug: gemcitabine hydrochloride — Given IV
  Other Names: gemcitabine; Gemzar; LY-188011

SUMMARY:
This phase I trial studies the side effects and best dose of ultrasound-guided photodynamic therapy with porfimer sodium when given together with gemcitabine hydrochloride in treating patients with locally advanced pancreatic cancer. Photodynamic therapy uses a drug, porfimer sodium, that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed. Drugs used in chemotherapy, such as gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving photodynamic therapy together with gemcitabine hydrochloride may be effect in patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of increasing porfimer sodium (PHO) dose and total energy by endoscopic ultrasound (EUS)-guided photodynamic therapy (PDT) for locally advanced unresectable pancreatic cancer (PC) in humans.

SECONDARY OBJECTIVES:

I. Quantify computed tomography (CT) detected volume of tumor necrosis produced by EUS-PDT.

II. Quantify rates of tumor size stabilization or decrease by EUS PDT and determine objective response rate per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.

III. Determine surgical downstaging off of abdominal vessels and resectability. IV. Determine changes in serum cancer antigen (CA) 19-9 levels with treatment. V. Evaluate progression-free and overall survival.

OUTLINE: This is a dose-escalation study of EUS-PDT with porfimer sodium.

Patients receive porfimer sodium intravenously (IV) on day 1 and undergo EUS-PDT on days 1, 3, 8, and 21. After completion of EUS-PDT, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 of courses 1 and 2 and on day 22 of courses 3 and 5. During courses 1-5, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. After course 5, treatment with gemcitabine hydrochloride repeats every 2 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, locally advanced measurable (at least bidirectional) adenocarcinoma of the pancreas (regardless of site) proven by biopsy or cytology and confirmed by surgical consultation
* Informed consent and authorization for the release of health information signed by the patient
* Karnofsky performance status >= 70%
* Life expectancy >= 3 months
* Females of childbearing potential and males must use an effective method of contraception

Exclusion Criteria:

* Metastatic (stage IV) disease (including involvement of the colon, adrenals, or kidney, or radiographic evidence of peritoneal seeding or pulmonary metastases)
* Previous chemotherapy, radiotherapy of other treatment for PC
* Gastric or duodenal wall invasion by the primary PC as assessed by CT or MRI and EUS staging
* Gastric or duodenal ulcer (at least 10 mm in size) within 10 mm of expected endoscopy puncture site(s) for PDT
* Esophageal or gastric varices
* Cystic component >= 25% the total volume of the tumor
* Ascites detected by CT, ultrasound (US) or MRI; (trace ascites will not be an exclusion)
* Bulky celiac adenopathy (i.e., >= 2.5 cm in diameter)
* Diagnosis of islet cell tumor, lymphoma, metastatic lesion, acinar cell (or other atypical pathologic malignancy)
* History of other malignancy in the past 2 years except carcinoma in situ of the cervix or bladder, non-melanomatous skin cancer or localized/early stage prostate cancer
* Unable to receive or previously intolerant of moderate and/or deep sedation
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) >= 3 x upper limit of normal (ULN)
* Total bilirubin >= 3 x ULN
* Alkaline phosphatase >= 3 x ULN
* International normalized ratio (INR) >= 1.5
* Partial thromboplastin time (PTT) ratio >= 1.5
* Serum creatinine >= 2.0 mg/dL
* Hematocrit =< 28% or hemoglobin =< 9 g/dL, but may have red blood cell (RBC) transfusion
* Platelet count =< 100,000/microliter (uL)
* Absolute neutrophil count (ANC) =< 1500/uL
* Clinically significant pancreatitis within 12 weeks of treatment with protocol therapy
* Contraindication to EUS-guided needle puncture into the pancreas
* History of coagulopathy or known thrombophilias
* Use of anticoagulants that cannot be discontinued both 5 days before and 5 days after EUS
* Clinical evidence of active infection of any type, including hepatitis B or C virus
* Pregnant or lactating women
* Experimental medications within the last 4 weeks prior to day 1
* Any surgery (including diagnostic laparoscopy and/or biliary +/- duodenal palliative bypass for inoperable PC) within the 2 weeks prior to day 1 of study protocol
* Chronic systemic corticosteroid use at superphysiologic doses (>= 10 mg prednisone per day or equivalent)
* Inability to avoid exposure of skin or eyes to direct sunlight or bright indoor light for at least 30 days
* Porphyria
* Inability to obtain venous access in the antecubital region to administer PHO or sedation for endoscopy procedures
* Significant concurrent medical or psychiatric illness which, in the opinion of the principal investigator would interfere with trial participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2013-04-19 (Actual); Primary Completion 2017-07-13 (Actual); Study Completion 2018-10-28 (Actual)

PRIMARY OUTCOMES:
Evaluate the number of subjects with adverse events which occur when up to 3 sites within the pancreas are treated with PDT using a total dose of 50 or 100 J per site | Up to 4 years
  Adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.0 which uses a scale of 1 (mild) to 5 (caused death).

SECONDARY OUTCOMES:
CT- or MRI-detected volume of tumor necrosis | Week 2
  Will be compared using paired t-tests or Wilcoxon rank sum tests as appropriate and changes will be plotted by maximal total energy of treatment to explore for dose-response effects.
Rates of tumor size stabilization or decease by EUS-PDT | Up to 4 years
  Will be compared using paired t-tests or Wilcoxon rank sum tests as appropriate and changes will be plotted by maximal total energy of treatment to explore for dose-response effects.
Objective response rate per RECIST | Up to 4 years
Surgical downstaging off of abdominal vessels or change in tumor unresectability | Up to 4 years
Change in CA 19-9 levels | Baseline to up to 4 years
  Will be compared using paired t-tests or Wilcoxon rank sum tests as appropriate and changes will be plotted by maximal total energy of treatment to explore for dose-response effects.
Progression-free survival | From the date of initial treatment to the earliest date of disease progression, resection of measurable tumor or death for patients who fail; and to the date of disease evaluation for patients who remain at risk for failure, assessed up to 4 years
  A Kaplan-Meier plot will be produced.
Overall survival | From the day of first treatment to the earlier of death (from any cause) and the last date of patient contact, assessed up to 4 years
  A Kaplan-Meier plot will be produced.

CONTACTS AND LOCATIONS:
Overall Officials: John M DeWitt, MD, Principal Investigator — Indiana University
Locations (1):
- IU Simon Cancer Center, Indianapolis, Indiana, United States

REFERENCES:
- [Derived] DeWitt JM, Sandrasegaran K, O'Neil B, House MG, Zyromski NJ, Sehdev A, Perkins SM, Flynn J, McCranor L, Shahda S. Phase 1 study of EUS-guided photodynamic therapy for locally advanced pancreatic cancer. Gastrointest Endosc. 2019 Feb;89(2):390-398. doi: 10.1016/j.gie.2018.09.007. Epub 2018 Sep 14. PMID 30222972